CLINICAL TRIAL: NCT01545089
Title: Use of a Fabric Mattress Cover for Patient Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: LOCAL/2011/LD-02; 2011-A01595-36 (Other: RCB number)
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Patient Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mattress protector days 1,2 (Experimental): A mattress protector is placed in the bed for the first two days and then removed for days 3 and 4.
  Interventions: Other: Mattress protector for days 1 and 2
- Mattress protector days 3,4 (Experimental): A mattress protector is not placed in the bed for the first two days and then added to the bed for days 3 and 4.
  Interventions: Other: Mattress protector for days 3 and 4

INTERVENTIONS:
Other: Mattress protector for days 1 and 2 — A mattress protector is placed in the bed for the first two days and then removed for days 3 and 4.
  Arms: Mattress protector days 1,2
Other: Mattress protector for days 3 and 4 — A mattress protector is not placed in the bed for the first two days and then added to the bed for days 3 and 4.
  Arms: Mattress protector days 3,4

SUMMARY:
The main objective of this research project is to measure the impact on patient satisfaction of the use of a fabric mattress cover fabric on a bedsheet protecting a plastic mattress.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has a planned hospitalization > 4 days
* The patient is "movable" within 48 hours

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Visual analog scale for patient comfort | 2 days
  score ranging from 0 to 10
Visual analog scale for patient comfort | 4 days
  score ranging from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Luc Duwig, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France